CLINICAL TRIAL: NCT03023449
Title: Diffuse Optical Monitoring With Inhaled Nitric Oxide
Acronym: DOMINO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Steven Messe (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor-Investigator, Steven Messe, Associate Professor of Neurology, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 824559
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Nitric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Controls (Experimental): The protocol will be a 35-minute monitoring session, during which cerebral hemodynamics will be monitored with both DCS and TCD, while blood pressure, heart rate, cardiac output, respiratory rate, end oxygen saturation, and inhaled nitric oxide concentration, are continuously monitored. 5 minutes of baseline hemodynamics will be assessed, after which the subject will breath iNO for 5 minutes, followed by 5 minutes of room air. This iNO/room air cycle will be repeated with a total of 3 different iNO concentrations. The full protocol will require 35 minutes. Subjects will be called at 24 hours after the monitoring session to determine any tolerability issues or adverse events.
  Interventions: Drug: Nitric Oxide
- Acute Ischemic Stroke (Experimental): Patients will be enrolled in the study within 72 hours of stroke symptom onset. The protocol will be a 35-minute monitoring session, during which cerebral hemodynamics will be monitored with both DCS and TCD, while blood pressure, heart rate, cardiac output, respiratory rate, end oxygen saturation, and inhaled nitric oxide concentration, are continuously monitored. 5 minutes of baseline hemodynamics will be assessed, after which the subject will breath iNO for 5 minutes, followed by 5 minutes of room air. This iNO/room air cycle will be repeated with a total of 3 different iNO concentrations. The full protocol will require 35 minutes. Subjects will be undergo a final assessment at 24 hours after the monitoring session to determine any tolerability issues or adverse events.
  Interventions: Drug: Nitric Oxide

INTERVENTIONS:
Drug: Nitric Oxide — Inhaled Nitric Oxide gas
  Other Names: iNO; NO2

SUMMARY:
This study is a non-randomized, Phase 2 clinical trial designed to measure the cerebral blood flow (CBF) response to inhaled nitric oxide in acute ischemic stroke patients and healthy subjects. The monitoring is a 35 minute session during which cerebral hemodynamics will be monitored with both diffuse correlation spectroscopy (DCS) and transcranial doppler ultrasonography (TCD) while blood pressure, heart rate, cardiac output, respiratory rate, end oxygen saturation, and inhaled nitric oxide (NO)/nitrogen dioxide (NO2) concentration, are continuously monitored.

ELIGIBILITY:
Inclusion Criteria:

Stroke Patients:

1. Age greater than 18
2. Acute ischemic stroke in the territory of the anterior, middle, or posterior cerebral artery, on either side of the brain
3. Study can be initiated within 72 hours of stroke symptom onset

3. Ability and willingness to sign informed consent

Healthy subjects:

1. Age greater than 18
2. Ability and willingness to sign informed consent

Exclusion Criteria:

Stroke subjects:

1. History of prior stroke or transient ischemic attack
2. Known cerebrovascular abnormality
3. History of congestive heart failure
4. Presence of pneumonia or active pulmonary infection
5. Current use of any NO donor medication (sodium nitroprusside or nitroglycerin)
6. Age less than 18 years
7. Skull defect that would interfere with CBF monitoring
8. Pregnancy
9. Structural brain lesion
10. Prior neurosurgical procedure
11. History of psychiatric disease
12. Any medical condition that the clinical investigator feels would pose a hazard to the subject if he/she participated in the study

Healthy subjects:

1. History of any neurological disease
2. History of stroke or transient ischemic attack
3. Known cerebrovascular abnormality
4. History of congestive heart failure
5. History of chronic pulmonary disease such as asthma or chronic obstructive pulmonary disease
6. Presence of pneumonia or active pulmonary infection
7. Current use of any NO donor medication (sodium nitroprusside or nitroglycerin)
8. Age less than 18 years
9. Skull defect that would interfere with CBF monitoring
10. Pregnancy (urine or blood tests will not be performed)
11. Structural brain lesion
12. Prior neurosurgical procedure
13. History of psychiatric disease
14. Any medical condition that the clinical investigator feels would pose a hazard to the subject if he/she participated in the study
15. Cognitive impairment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-04-04 (Actual); Primary Completion 2021-03-21 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in cerebral blood flow during the administration of iNO | Conclusion of the 35 minute protocol

SECONDARY OUTCOMES:
Change in blood flow velocity as measured by TCD during iNO administration | Conclusion of the 35 minute protocol
Change in mean arterial blood pressure (MAP) during iNO administration | Conclusion of the 35 minute protocol
Time to maximum CBF effect after the introduction of iNO | Conclusion of the 35 minute protocol
Duration of residual effect after cessation of iNO (time to return to baseline) | Conclusion of the 35 minute protocol

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Messe, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No